CLINICAL TRIAL: NCT00031707
Title: Phase III Double-Blind, Placebo-Controlled Randomized Comparison of Megestrol Acetate (Megace) Versus an N-3 Fatty Acid (EPA) Enriched Nutritional Supplement Versus Both for the Treatment of Cancer Cachexia and Anorexia
Brief Title: Comparison of Megestrol and/or Omega-3 Fatty Acid-Enriched Nutritional Supplement in Treating Patients With Cancer-Related Weight Loss and Lack of Appetite
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-989255; CDR0000069218 (Registry Identifier: PDQ (Physician Data Query)); CAN-NCIC-SC18; NCI-P02-0205
Record Dates: First submitted 2002-03-08; First posted 2003-08-05 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Anorexia; Cachexia
Keywords: anorexia; cachexia
MeSH Terms: conditions — Anorexia; Cachexia | interventions — Eicosapentaenoic Acid; Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- megestrol + placebo (Active Comparator): Patients receive oral megestrol once daily and oral placebo twice daily. Treatment continues in the absence of unacceptable toxicity and as long as the patient and physician feel it is beneficial.
  Quality of life is assessed at baseline, weekly for 1 month, and then monthly thereafter during study treatment.
  Patients are followed every 6 months for 5 years.
  Interventions: Drug: megestrol acetate; Other: placebo
- eicosapentaenoic acid + placebo (Active Comparator): Patients receive oral placebo once daily and an eicosapentaenoic acid (EPA)-enriched nutritional supplement twice daily. Treatment continues in the absence of unacceptable toxicity and as long as the patient and physician feel it is beneficial.
  Quality of life is assessed at baseline, weekly for 1 month, and then monthly thereafter during study treatment.
  Patients are followed every 6 months for 5 years.
  Interventions: Dietary Supplement: eicosapentaenoic acid; Other: placebo
- megestrol + eicosapentaenoic acid (Experimental): Patients receive oral megestrol once daily and an EPA-enriched nutritional supplement twice daily. Treatment continues in the absence of unacceptable toxicity and as long as the patient and physician feel it is beneficial.
  Quality of life is assessed at baseline, weekly for 1 month, and then monthly thereafter during study treatment.
  Patients are followed every 6 months for 5 years.
  Interventions: Dietary Supplement: eicosapentaenoic acid; Drug: megestrol acetate

INTERVENTIONS:
Dietary Supplement: eicosapentaenoic acid
  Arms: eicosapentaenoic acid + placebo; megestrol + eicosapentaenoic acid
Drug: megestrol acetate
  Arms: megestrol + eicosapentaenoic acid; megestrol + placebo
Other: placebo
  Arms: eicosapentaenoic acid + placebo; megestrol + placebo

SUMMARY:
RATIONALE: Megestrol and /or an omega-3 fatty acid-enriched nutritional supplement may improve cancer-related weight loss and lack of appetite. It is not yet known whether megestrol alone, an omega-3 fatty acid-enriched nutritional supplement alone, or a combination of both is most effective in treating cancer-related weight loss and loss of appetite.

PURPOSE: Randomized phase III trial to compare the effectiveness of megestrol with or without an omega-3 fatty acid-enriched nutritional supplement to that of the omega-3 fatty acid-enriched nutritional supplement alone in treating patients who have cancer-related weight loss and lack of appetite.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the appetite-stimulating properties of megestrol vs an eicosapentaenoic acid-enriched nutritional supplement vs both, in terms of patient weight, rate of weight change, and appetite, in patients with cancer-related cachexia and anorexia.
* Determine the effect of these regimens on nausea and vomiting in these patients.
* Assess quality of life in patients treated with these regimens.
* Determine the toxic effects of these regimens in these patients.
* Compare overall survival of patients treated with these regimens.
* Correlate interleukin-6 concentration changes with appetite and weight changes in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to primary cancer (lung vs gastrointestinal vs other), severity of weight loss in the past 2 months (less than 10 pounds vs 10 pounds or more), planned concurrent chemotherapy (yes vs no), age (under 50 vs 50 and over), and prognosis (good vs bad vs unsure). Patients are randomized to 1 of 3 treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven cancer other than brain, breast, ovarian, endometrial, or prostate cancer

  * Compelling clinical evidence of cancer is allowed when tissue sample is unobtainable
* Considered incurable with available therapies
* At least 5 pounds weight loss within the past 2 months (excluding perioperative weight loss) and/or have estimated caloric intake of less than 20 cal/kg daily
* Weight loss must be perceived as a problem by the patient
* Potential weight gain must be considered beneficial by the attending physician
* No history of primary brain cancer or brain metastases
* No clinical evidence of ascites

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Cardiovascular:

* No poorly controlled congestive heart failure
* No poorly controlled hypertension
* No history of thromboembolic disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Alert and mentally competent
* Able to reliably take oral medication
* No known mechanical obstruction of the alimentary tract, malabsorption, or intractable vomiting (more than 5 episodes per week)
* No diabetes requiring insulin
* Diabetes requiring an oral hypoglycemic agent or diet control allowed

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* Concurrent chemotherapy allowed

Endocrine therapy:

* At least 1 month since prior adrenal steroids, androgens, progestational agents, or appetite stimulants (e.g., dronabinol)
* No concurrent adrenal steroids, androgens, other progestational agents, or appetite stimulants (e.g., dronabinol)

  * Inhalant, topical, or optical steroids allowed
  * Short-term dexamethasone as an anti-emetic during chemotherapy allowed

Radiotherapy:

* Concurrent radiotherapy allowed

Other:

* No tube feedings or parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2000-03; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Compare the appetite-stimulating properties (eg, patient weight, rate of weight change, and appetite) | Up to 5 years

SECONDARY OUTCOMES:
Assess quality of life | Up to 5 years
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (44):
- United States (22):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Canada (22):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Nanaimo Cancer Clinic, Nanaimo, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - William Osler Health Centre, Brampton, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Result] Jatoi A, Rowland K, Loprinzi CL, Sloan JA, Dakhil SR, MacDonald N, Gagnon B, Novotny PJ, Mailliard JA, Bushey TI, Nair S, Christensen B; North Central Cancer Treatment Group. An eicosapentaenoic acid supplement versus megestrol acetate versus both for patients with cancer-associated wasting: a North Central Cancer Treatment Group and National Cancer Institute of Canada collaborative effort. J Clin Oncol. 2004 Jun 15;22(12):2469-76. doi: 10.1200/JCO.2004.06.024. PMID 15197210